CLINICAL TRIAL: NCT00832039
Title: Prospective, Randomized Multicenter Trial of Adjunctive Intravenous Therapy With Sodium-selenite(Selenase®, Double-blinded) and a Procalcitonin Guided Causal Therapy (Open) of Severe Sepsis or Septic Shock.
Brief Title: Placebo Controlled Trial of Sodium Selenite and Procalcitonin Guided Antimicrobial Therapy in Severe Sepsis
Acronym: SISPCT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kompetenznetz Sepsis (Network)
Collaborators: Biosyn (Industry); Brahms AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: EudraCT 2007-004333-42; 01 KI 01 06 (Other Grant/Funding Number: bmbf); SE120301S (Other: Biosyn)
Record Dates: First submitted 2009-01-28; First posted 2009-01-29 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Severe Sepsis; Septic Shock
Keywords: sepsis; adjunctive therapy; sodium-selenite; procalcitonin
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Selenious Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- SelPCT (Active Comparator): Patient receives sodium-selenite; causal therapy is guided by a PCT based algorithm.
  Interventions: Drug: sodium-selenite; Procedure: Procalcitonin guided therapy
- SelKon (Active Comparator): Patient receives sodium-selenite; causal therapy is not guided by a PCT based algorithm.
  Interventions: Drug: sodium-selenite
- PlacPCT (Placebo Comparator): Patient receives placebo; causal therapy is guided by a PCT based algorithm.
  Interventions: Drug: Placebo; Procedure: Procalcitonin guided therapy
- PlacKon (Placebo Comparator): Patient receives placebo; causal therapy is not guided by a PCT based algorithm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: sodium-selenite — An intravenous bolus of 1000 µg followed by a continuous intravenous infusion of 1000 µg/day until patient is discharged from the ICU but not more than 21 applications à 24 hours.
  Other Names: selenase T
  Arms: SelKon; SelPCT
Drug: Placebo — An intravenous bolus of placebo followed by a continuous intravenous infusion with placebo until patient is discharged from the ICU but not more than 21 applications à 24 hours.
  Other Names: 0.9 % sodium chlorid
  Arms: PlacKon; PlacPCT
Procedure: Procalcitonin guided therapy — Causal therapy of sepsis is guided by applying the following algorithm:
  Day 4: PCT drop from baseline >=50%: no change in causal therapy; PCT drop from baseline <50%: change or optimize antimicrobial therapy, new intervention (i.e. surgery, diagnostics) recommended for source control.
  Day 7, 10, 14: PCT <=1.0 ng/ml: finish antimicrobial therapy; PCT >1.0 ng/ml and PCT drop from last PCT measurement >=50%: finish antimicrobial therapy; PCT >1.0 ng/ml and PCT drop from last PCT measurement <50%: change or optimize antimicrobial therapy, new intervention (i.e. surgery, diagnostics) recommended for source control.
  Arms: PlacPCT; SelPCT

SUMMARY:
Severe sepsis and septic shock are diseases of infectious origin with a high risk of death. The purpose of this study is to determine whether the intravenous application of selenium (given as sodium-selenite) can reduce mortality in patients with severe sepsis or septic shock. Additionally, it is investigated, whether the measurement of procalcitonin - a marker of infection - can be used to guide anti-infectious measures in this disease.

DETAILED DESCRIPTION:
This is a multicenter trial of the German Network Sepsis (SepNet) on patients with severe sepsis or septic shock. This study is supported by unrestricted grants.

The release of reactive oxygen species is an important factor in the development of sepsis induced multiorgan dysfunction syndrome. Common protection mechanisms are impaired in this syndrome. Serum levels of selenium, a cofactor of the glutathionperoxidase, are reduced. Several studies suggest a benefit of selenium application in patients with severe sepsis but data from large clinical trials are not available. After inclusion into the study, patients are randomly allocated to a placebo or selenium group. Treating physicians and patients are blinded regarding the allocation. The selenium group receives sodium selenite intravenously - 1000 µg as a bolus followed by a continuous infusion of 1000 µg per day until the end of ICU treatment but not longer than 21 days.

Procalcitonin (PCT) is a biomarker which is elevated in the blood of patients with severe sepsis/septic shock. Data from patients with community acquired pneumonia demonstrated that this biomarker can be used to decide on the duration of antimicrobial therapy. Studies with small sample size seem to confirm this in ICU patients with severe sepsis. However, this needs to be confirmed in a larger cohort. All patients are randomly allocated to a PCT guided algorithm or a control group. In the PCT-guided group, PCT is measured at randomization, day 4, 7, 10, and 14. Depending on the PCT course, the protocol recommends to change, alter, or stop anti-infectious measures. In the control group, anti-infectious therapy is left to the discretion of the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Severe sepsis or septic shock according to ACCP/SCCM criteria
* Onset of severe sepsis or septic shock <24 h
* Age >= 18 years
* Informed consent

Exclusion Criteria:

* Pregnant or breast-feeding women
* Fertile female women without effective contraception
* Participation in interventional clinical trial within the last 30 days
* Current participation in any study
* Former participation in this trial
* Selenium intoxication
* No commitment to full patient support (i.e. DNR order)
* Patient's death is considered imminent due to coexisting disease
* Relationship of the patient to study team member (i.e. colleague, relative)
* Infection where guidelines recommend a longer duration of antimicrobial therapy (i.e. endocarditis, tuberculosis, malaria etc)
* Immunocompromised patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1089 (Actual)
Dates: Start 2009-11; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 28 days

SECONDARY OUTCOMES:
Mean total SOFA and SOFA subscores | study duration
All cause mortality | 90 days
Frequency and duration of mechanical ventilation | 90 days
Frequency and duration of vasopressor support | 90 days
Frequency of adverse events and severe adverse events | study duration
Clinical cure and microbiological cure | days 4, 7, 10, 14
Duration of antimicrobial therapy | study duration
Costs of antimicrobial therapy | study duration
Time to change of antibiotic therapy | duration of study
Days alive without antimicrobial therapy | study duration
Frequency of resistancies against antibiotics (VRE, MRSA, ESBL) | study duration
ICU length of stay | 90 days
Hospital length of stay | 90 days
Rate of surgical procedures for focus control | study duration
Rate of procedures to diagnose infections | study duration
Frequency of new infections | study duration

CONTACTS AND LOCATIONS:
Overall Officials: Konrad Reinhart, M.D., Study Chair — University Hospital Jena; Dep. of Anesthesiology and Intensive Care Medicine; Markus Löffler, Study Director — University Leipzig; Koordinierungszentrum für Klinische Studien Leipzig (KKSL); Thomas Deufel, M. D., Study Director — University Hopitel Jena, Institute for Medical Chemistry
Locations (35):
- Germany (35):
  - University Hospital Aachen - Dep. of Intensive Care Medicine, Aachen
  - Klinikum Augsburg - Dep. of Anesthesiology and Intensive Care Medicine, Augsburg
  - Klinikum Augsburg - Dep. of Medicine I, Augsburg
  - Military Hospital Berlin - Dep. of Anaesthesiology and Intensive Care Medicine, Berlin
  - Charité Berlin - Dep. of Anesthesiology and Intensive Care Medicine, Berlin
  - Vivantes Klinikum Neukölln - Dep. of Anesthesiology, Intensive Care Medicine and Pain Therapy, Berlin
  - DRK-Kliniken Berlin-Köpenick - Dep. of Anesthesiology, Pain Therapy, and Intensive Care Medicine, Berlin
  - Charité Berlin - Campus Virchow-Klinikum - Dep. of Nephrology, Berlin
  - Ev. Krankenhaus Gilead - Dep. of Anesthesiology, Bielefeld
  - University Hospital Bonn - Dep. of Anesthesiology and Intensive Care Medicine, Bonn
  - University Hospital Köln - Dep. of Medicine I, Cologne
  - Krankenhaus Dresden-Friedrichstadt, Dresden
  - University Hospital Dresden - Dep. of Anesthesiology and Intensive Care Med., Dresden
  - HELIOS Klinikum Erfurt - Dep. of Anesthesiology and Intensive Care Medicine, Erfurt
  - University Erlangen-Nürnberg - Dep. of Medicine IV, Erlangen
  - J.-W. Goethe University Hospital - Dep. of Anaesthesiology, Intensive Care Medicine and Pain Therapy, Frankfurt am Main
  - University Hospital Freiburg- Dep. of Surgery, Freiburg im Breisgau
  - Georg August Universität Göttingen - Dep. of Anesthesiology and Intensive Care Medicine, Göttingen
  - Ernst-Moritz-Arndt-Universität Greifswald - Dep. of Anesthesiology and Intensive Care Medicine, Greifswald
  - Martin-Luther-Universität Halle-Wittenberg - Dep. of Anesthesiology, Halle
  - University Hospital Halle - Dep. of Medicine III, Halle
  - Universitätsklinikum Hamburg-Eppendorf - Dep. of Intensive Care Medicine, Hamburg
  - Westküstenklinikum Heide - Dep. of Anesthesiology and Intensive Care Medicine, Heide
  - University Hospital Heidelberg - study center Anesthesiology/Surgery, Heidelberg
  - University Hospital Jena, Dep. of Anesthesiology and Intensive Care Medicine, Jena
  - University Hospital Kiel - Dep. of. Anesthesiology and Intensive Care Medicine, Kiel
  - St. Elisabeth-Krankenhaus - Dep. of Anesthesiology, Köln-Hohenlind
  - University Hospital Leipzig - Dep. of Anesthesiology and Intensive Care Medicine, Leipzig
  - University Hospital Mannheim - Dep. of Medicine I, Mannheim
  - University Hospital Munich - Dep. of Internal Medicine, Munich
  - University Hospital Munich - Dep. of Anaesthesiology, Munich
  - Hospital Munich Harlaching - Dep. of Internal Acute Medicine and Prevention, Munich
  - Krankenhaus München-Neuperlach - Dep. of Anesthesiology, München
  - University Hospital Münster - Dep. of Anesthesiology and Intensive Care Medicine, Münster
  - Klinikum Oldenburg GmbH - Dep. of Anesthesiology, Oldenburg

REFERENCES:
- [Result] Bloos F, Trips E, Nierhaus A, Briegel J, Heyland DK, Jaschinski U, Moerer O, Weyland A, Marx G, Grundling M, Kluge S, Kaufmann I, Ott K, Quintel M, Jelschen F, Meybohm P, Rademacher S, Meier-Hellmann A, Utzolino S, Kaisers UX, Putensen C, Elke G, Ragaller M, Gerlach H, Ludewig K, Kiehntopf M, Bogatsch H, Engel C, Brunkhorst FM, Loeffler M, Reinhart K; for SepNet Critical Care Trials Group. Effect of Sodium Selenite Administration and Procalcitonin-Guided Therapy on Mortality in Patients With Severe Sepsis or Septic Shock: A Randomized Clinical Trial. JAMA Intern Med. 2016 Sep 1;176(9):1266-76. doi: 10.1001/jamainternmed.2016.2514. PMID 27428731
- [Derived] Guo A, Srinath J, Feuerecker M, Crucian B, Briegel J, Boulesteix AL, Kaufmann I, Chouker A. Immune function testing in sepsis patients receiving sodium selenite. J Crit Care. 2019 Aug;52:208-212. doi: 10.1016/j.jcrc.2019.05.001. Epub 2019 May 4. PMID 31102938
- [Derived] Feuerecker M, Sudhoff L, Crucian B, Pagel JI, Sams C, Strewe C, Guo A, Schelling G, Briegel J, Kaufmann I, Chouker A. Early immune anergy towards recall antigens and mitogens in patients at onset of septic shock. Sci Rep. 2018 Jan 29;8(1):1754. doi: 10.1038/s41598-018-19976-w. PMID 29379043
- See also: German Sepsis Society — http://www.sepsis-gesellschaft.de
- See also: Competence Network Sepsis (SepNet) — http://www.sepsis-gesellschaft.de/DSG/Deutsch/SepNet?sid=nbGlH39rI6b9u2fBVVhxiM&iid=1
- See also: Surviving Sepsis Campaign — http://www.survivingsepsis.org